CLINICAL TRIAL: NCT01631071
Title: Open, Non-randomized Trial to Assess the Immunogenicity and Safety of the 2012/2013-Season Virosomal Subunit Influenza Vaccine in Elderly and Young Subjects According to EMA Regulations
Brief Title: Re-licensing Study to Assess Virosomal Influenza Vaccine Formulated With WHO Recommended Influenza Strains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ADD-V-A003
Record Dates: First submitted 2012-06-25; First posted 2012-06-28 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-02

CONDITIONS: Influenza
Keywords: Influenza; Virus; Vaccination; Virosomal influenza vaccine
MeSH Terms: conditions — Influenza, Human; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elderly subjects aged over 60 years (Experimental)
  Interventions: Biological: Virosomal influenza vaccine
- Adults from 18 to 60 years old inclusive (Experimental)
  Interventions: Biological: Virosomal influenza vaccine

INTERVENTIONS:
Biological: Virosomal influenza vaccine — Intramuscular administration (M. deltoideus) of a single dose of 0.5 mL virosomal influenza vaccine

SUMMARY:
The study is to assess whether the virosomal influenza vaccine for season 2012/2013 fulfills the EMA requirements for re-registration of influenza vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male adults aged ≥18 on Day 1
* Written informed consent
* Female subjects of childbearing potential using and willing to continue using an acceptable method of contraception unless surgically sterilized/hysterectomized or post-menopausal for more than 2 years

Exclusion Criteria:

* Acute exacerbation of bronchopulmonary infection (cough, sputum, lung findings) or other acute disease
* Acute febrile illness (≥38.0 °C)
* Prior vaccination with an influenza vaccine in the past 330 days
* Known hypersensitivity to any vaccine component
* Previous history of a serious adverse reaction to influenza vaccine
* History of egg protein allergy or severe atopy
* Known blood coagulation disorder
* Chronic (longer than 14 days) administration of immunosuppressants or other immune-modifying drugs within 6 months before the first dose of the study vaccine, including oral corticosteroids in dosages of ≥0.5 mg/kg/d prednisolone or equivalent (inhaled or topical steroids are allowed)
* Known immunodeficiency (incl. leukemia, HIV seropositivity), cancer
* Investigational medicinal product received in the past 3 months (90 days) starting from the first day of the month following the last visit in a previous study
* Treatment with immunoglobulins or blood transfusion(s) received in the past 3 months (90 days)
* Pregnancy or lactation
* Participation in another clinical trial
* Employee at the investigational site, or relative of the investigator
* Subjects who in the view of the investigator will not comply with study procedures and/or visit requirements as per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — CROSS-Research SA
Locations (1):
- CROSS-Research SA, Arzo, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 03 August 2012 to 27 August 2012; outpatient study
Period: Overall Study
Arm/Group | Elderly Subjects Aged Over 60 Years | Adults From 18 to 60 Years Old Inclusive
Started | 55 | 55
Completed | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elderly Subjects Aged Over 60 Years | Adults From 18 to 60 Years Old Inclusive | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 55 | 78
  >=65 years | 32 | 0 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (4.42) | 41.0 (11.52) | 53.6 (15.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 64
  Male | 21 | 25 | 46
Region of Enrollment [Number; unit: participants]
  Switzerland | 55 | 55 | 110

OUTCOME MEASURES:

1. Primary Outcome: Seroprotection
Description: Seroprotection rate, defined as proportion of subjects with HI antibody titer ≥1:40 (The primary endpoints are the immunogenicity parameters for HA assessed via hemagglutinin inhibition method (HI). These parameters were analyzed according to the EMA "Note for guidance on harmonisation of requirements for influenza vaccines," 1997)
Time Frame: Day 22 +/- 2 days
Population: Intent-to-treat, vaccinated subjects with available pre- and post-vaccination titers
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Elderly Subjects Aged Over 60 Years | Adults From 18 to 60 Years Old Inclusive
Number analyzed (Participants) | 55 | 55
percentage of subjects
  Percentage seroprotected subjects: A/H1N1 | 94.5 [84.9 to 98.9] | 100 [93.5 to 100]
  Percentage seroprotected subjects: A/H3N2 | 100 [93.5 to 100] | 100 [93.5 to 100]
  Percentage seroprotected subjects: B strain | 100 [93.5 to 100] | 100 [93.5 to 100]

2. Secondary Outcome: Number of Participants With Local and Systemic Adverse Events, as a Measure of Safety and Tolerability
Description: Solicited local and systemic AEs, Unsolicited AEs
  Unsolicited AEs were collected from baseline (Day 1) to 3 weeks after vaccination (Day 22 ± 2 days).
  Solicited local and systemic AEs were collected by subjects diary from Day 1 (day of vaccination) to Day 4
Time Frame: Baseline (Day 1) and 3 weeks after vaccination (Day 22 ± 2 days)
Measure: Number; unit: participants
Arm/Group | Elderly Subjects Aged Over 60 Years | Adults From 18 to 60 Years Old Inclusive
Number analyzed (Participants) | 55 | 55
participants
  AEs (unsolicited and unsolicited) | 23 | 32
  Unsolicited AEs | 4 | 5
  Solicited local AEs | 20 | 30
  Solicited systemic AEs | 1 | 7

3. Primary Outcome: Seroconversion
Description: Seroconversion rate, defined as proportion of subjects with ≥4-fold increase in HI antibody titer and with a titer of ≥1:40 (The primary endpoints are the immunogenicity parameters for HA assessed via hemagglutinin inhibition method (HI). These parameters were analyzed according to the EMA "Note for guidance on harmonisation of requirements for influenza vaccines," 1997)
Time Frame: Day 22 +/- 2 days
Population: Intent-to-treat, vaccinated subjects with available pre- and post-vaccination titers
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Elderly Subjects Aged Over 60 Years | Adults From 18 to 60 Years Old Inclusive
Number analyzed (Participants) | 55 | 55
percentage of subjects
  Percentage seroconverted subjects: A/H1N1 | 43.6 [30.3 to 57.7] | 58.2 [44.1 to 71.3]
  Percentage seroconverted subjects: A/H3N2 | 27.3 [16.1 to 41.0] | 36.4 [23.8 to 50.4]
  Percentage seroconverted subjects: B strain | 34.5 [22.2 to 48.6] | 43.6 [30.3 to 57.7]

4. Primary Outcome: Geometric Mean Titer
Description: GMT of HI antibodies and fold-increase in GMT (The primary endpoints are the immunogenicity parameters for HA assessed via hemagglutinin inhibition method (HI). These parameters were analyzed according to the EMA "Note for guidance on harmonisation of requirements for influenza vaccines," 1997)
Time Frame: Day 22 +/- 2 days
Population: Intent-to-treat, vaccinated subjects with available pre- and post-vaccination titers
Measure: Number (95% Confidence Interval); unit: GMT fold increase from baseline
Arm/Group | Elderly Subjects Aged Over 60 Years | Adults From 18 to 60 Years Old Inclusive
Number analyzed (Participants) | 55 | 55
GMT fold increase from baseline
  GMT fold increase: A/H1N1 | 4.25 [3.26 to 5.54] | 4.62 [3.48 to 6.15]
  GMT fold increase: A/H3N2 | 2.70 [2.18 to 3.33] | 2.78 [2.24 to 3.44]
  GMT fold increase: B strain | 2.78 [2.30 to 3.36] | 3.27 [2.59 to 4.13]

ADVERSE EVENTS:
Arm/Group | Elderly Subjects Aged Over 60 Years | Adults From 18 to 60 Years Old Inclusive
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 23/55 | 32/55
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elderly Subjects Aged Over 60 Years (N=55) | Adults From 18 to 60 Years Old Inclusive (N=55)
Malaise (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 9 (9) | 10 (10)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 7 (7) | 12 (12)
Injection site pain (General disorders) | 17 (17) | 28 (28)
Chills (shivering) (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 7 (7)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Material for public dissemination will be submitted to the Sponsor for review at least ninety (90) days prior to submission for publication, public dissemination, or review by a publication committee.